CLINICAL TRIAL: NCT06610396
Title: Ex Onc SLED: a Pilot Study Utilizing a Weighted Sled for Horizontal Resistance Training
Brief Title: Ex Onc SLED: a Study Utilizing a Weighted Sled for Horizontal Resistance Training
Status: Recruiting | Type: Observational
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Colin Champ, MD, Radiation Oncologist, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Other Study IDs: 2024-115-SG
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: exercise; resistance training
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This protocol seeks to analyze patient adherence and outcomes after monitored exercise sessions utilizing primarily weighted sled pushes and pulls for linearly progressed resistance training of individuals who have been diagnosed with cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-89 years
2. Women of child-bearing potential must verbally confirm lack of pregnancy prior to enrollment. They should also consent to use adequate contraception during the course of the study.
3. Participants must be determined capable of engaging in resistance training by exercise personnel and/or study PI and must be able to stand.
4. Participants must complete an assessment by EOC staff and be determined safe to engage in the workout regimen by the study exercise personnel. Any individuals not deemed safe to participate in the basic EOC exercise program will be referred to physical therapy or elsewhere

Exclusion Criteria:

1. Severe arthritic, joint, cardiovascular, or musculoskeletal condition that would interfere with exercise program
2. Individuals deemed able to engage in more intense resistance training utilizing compound movements will not be eligible
3. Pregnant women

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with cancer on an exercise program at the AHN Exercise Oncology and Resiliency Center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Change in Adipose Tissue (InBody, kg) | Baseline and study completion, up to 6 months.
  Change in adipose tissue (kg) pre and post resistance training regimen measured via InBody 970 bioelectrical impedance analysis
Change in Adipose Tissue (Ultrasound, Lbs) | Baseline and study completion, up to 6 months.
  Change in adipose tissue (pounds) pre and post resistance training regimen measured via ultrasound.
Change in Muscle Mass | Baseline and study completion, up to 6 months.
  Changes in percent muscle mass (measured by InBody bioelectrical impedance analysis) and percent fat-free mass (measured by ultrasound) from baseline to six months

SECONDARY OUTCOMES:
Intervention Compliance Rate during Exercise Program (Adherence) | Through study completion, up to 6 months.
  Percentage of exercise sessions attended by each participant
Feasibility of the Exercise Program | Through study completion, up to 6 months.
  Tracking of participant completion status.
Adverse Events (Safety) | Through study completion, up to 6 months.
Changes in Timed Up and Go Test Performance at baseline and post-exercise assessment | Baseline and study completion, up to 6 months.
  An individual stands from a chair, walks ten feet and back, and then sits down. This is timed and recorded in seconds.
Changes in Functional Mobility Score at baseline and post-exercise assessment | Baseline and study completion, up to 6 months.
  During the test, 7 movement patterns are assessed and each one is rated between 0 and 3 by an examiner. These movements include the deep squat, hurdle step, inline lunge, shoulder mobility test, active straight leg raise, trunk stability push up, and rotary stability test. A score of zero is given if any pain is felt during the movement, 1 if the subject is unable to perform the movement, 2 if the subject performs the movement through compensatory movements, and 3 if the movement is performed correctly. Each movement score is summed and a final score out of 21 is calculated. A score below 14 is felt to identify individuals at risk of injury.
Changes in Y-Balance Test Scores at baseline and post-exercise assessment | Baseline and study completion, up to 6 months.
  Reach distances in three directions (anterior, posteromedial, and posterolateral) measured in centimeters.
Changes in EuroQol-5 Dimensions (EQ-5D) at baseline and post-exercise assessment | Baseline assessment (prior to program) and at exercise program completion.
  EuroQol-5 Dimensions-5 Levels total score for the 5 questions ranges from 5 (no problems on any dimension) to 25 (extreme problems on all dimensions). This is calculated by assigning scores of 1 (minimum), 2, 3, 4, and 5 (maximum), to the response categories of "no problems", "slight problems", "moderate problems", "severe problems", and "extreme problems"/"unable to", respectively. Higher scores mean worse outcomes.
Changes in Patient Health Questionnaire-9 (PHQ9) depression score at baseline and post-exercise assessment | Baseline and study completion, up to 6 months.
  Patient Health Questionnaire-9 total score for the 9 questions ranges from 0 (no depression) to 27 (highest level of depression). This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum), to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. Higher scores mean a worse outcome.
Changes in General Anxiety Disorder-7 (GAD7) anxiety score at baseline and post-exercise assessment | Baseline and study completion, up to 6 months.
  General Anxiety Disorder-7 total score for the seven questions ranges from 0 (no anxiety) to 21 (highest level of anxiety). This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum), to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. Higher scores mean a worse outcome.
Changes in grip strength at baseline, throughout, and post- exercise assessment | Through study completion, up to 6 months.
  Assessed via a Jamar Hand Dynamometer Grip Strength Measurement Meter bilaterally at the neutral position and with the arm over the head
Changes in load lifted during sled exercises at baseline, throughout, and post- exercise assessment | Through study completion, up to 6 months.
  Maximum weight lifted during sled training
Changes in resting metabolic rate at baseline and post-exercise assessment | Through study completion, up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, MD, Principal Investigator — AHN Radiation Oncology
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States